CLINICAL TRIAL: NCT02941523
Title: Phase Ia/Ib and Potential Phase IIa Study of the Safety and Pharmacokinetics of NOX66 Both as a Monotherapy and in Combination With Carboplatin in Patients With Refractory Solid Tumours
Brief Title: Safety, PK and Efficacy of NOX66 as a Monotherapy and Combined With Carboplatin in Refractory Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NOX66-001A
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — phenoxodiol; Carboplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1a NOX66 (Experimental): NOX66 administered daily for 14 day in a 21-day treatment cycle. NOX66 treatment given to two cohorts of patients as 1 of 2 dose regimens:
  Regimen 1: 400 mg; Regimen 2: 800 mg (idronoxil)
  Interventions: Drug: NOX66
- 1b NOX66 and Carboplatin (combined) (Experimental): NOX66 administered on Days 1-7 and carboplatin IV infusion on Day 2 of each 28-day treatment cycle up to 6 cycles.
  NOX66 at the same dosage received in the Run-In Arm combined with 2 carboplatin doses starting with low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
  Interventions: Drug: NOX66; Drug: Carboplatin
- 2a NOX66 and Carboplatin (Experimental): This arm triggered by observed meaningful clinical responses from the 1b Combination Arm in particular disease indications.
  Treatment NOX66 + carboplatin administered over 6 cycles each of 28-days at observed clinical response dosage. A maximum of 2 cohorts, each comprising patients with specific tumour type.
  Interventions: Drug: NOX66; Drug: Carboplatin

INTERVENTIONS:
Drug: NOX66 — NOX66 administration
  Other Names: Idronoxil
Drug: Carboplatin — Carboplatin administration
  Other Names: Paraplatin
  Arms: 1b NOX66 and Carboplatin (combined); 2a NOX66 and Carboplatin

SUMMARY:
The study evaluates the safety and activity of NOX66 in patients with refractory solid tumors that are non responsive to standard therapies.

This is a two part with a potential third part, open-label, multicenter, dose escalation study of NOX66 as monotherapy and in combination with carboplatin.

DETAILED DESCRIPTION:
Idronoxil is a synthetic small molecule that pre-clinical studies have identified as a strong candidate for development as a chemo-sensitising drug.

Human studies using idronoxil administered in oral and intravenous dosage forms have shown that the drug is highly susceptible to Phase 2 metabolism, resulting in loss of bio-activity.

NOX66 is idronoxil in a new dosage formulation developed specifically to protect the drug from Phase 2 metabolism and thereby ensure retention of the majority of administered drug in a bio-active form.

The main purpose of the current study is to confirm the safety of the new dosage formula both as a monotherapy and in combination with carboplatin, given that it is anticipated that the drug will be present in the body in a bio-active form at considerably higher levels than previously achieved.

A secondary objective is to observe if NOX66 is able to restore response to carboplatin in tumours considered unresponsive to this chemotherapy, and moreover to provide a meaningful clinical benefit in combination with a lower-than-normal dosage of carboplatin.

Patients will be drawn from 5 cancer types: prostate cancer, lung cancer, breast cancer, ovarian cancer, head and neck cancer.

The study will commence with a Phase 1a (Run-in) arm comparing the relative tolerability and safety of two different dosages of idronoxil/NOX66 as a 14-day monotherapy course.

Providing there is no dose limiting toxicity (DLT), patients then progress onto the Phase 1b (Combination) arm of the study, remaining on the same dosage. In this arm, patients receive 6 treatment cycles, each of 28 days comprising NOX66 (idronoxil) treatment on Days 1-7 and carboplatin on Day 2 of each treatment cycle.

Any meaningful clinical responses occurring in the Phase 1b (Combination) Arm will trigger a Phase IIa (Combination) Arm where an additional 10 patients will be recruited into a maximum of 2 cohorts of the same tumour type (prostate, lung, breast, ovarian, or head and neck). These patients will receive the same combination dosage providing the observed clinical responses and treated with that dosage for a maximum of 6 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Male or female ≥18 years of age
3. Histologic or cytologic confirmed locally advanced or metastatic cancer that has no standard therapeutic alternatives.
4. ECOG Performance status 0-1
5. A minimum life expectancy of 12 weeks
6. Adequate bone marrow, hepatic and renal function as evidenced by:

   * Absolute neutrophil count (ANC) > 1.5 x 109/L
   * Platelet count > 100 x 109/L
   * Hemoglobin > 9.0 g/dL
   * Serum bilirubin < 1.5 x ULN
   * AST/ALT (SGOT/SGPT) 2.5 x ULN for the reference laboratory or < 5 x ULN in the presence of liver metastases
   * Serum creatinine 1.5 x ULN
7. Female patients who are known to be capable of conception should have a negative serum pregnancy test (beta-human chorionic gonadotropin (β-hCG)) within 1 week of starting the study
8. All potentially fertile patients will agree to use an effective form of contraception during the study and for 90 days following the last dose of NOX66 (an effective form of contraception is defined as an oral contraceptive or a double barrier method
9. At least 4 weeks must have elapsed prior to commencement of NOX66 treatment since prior chemotherapy, investigational drug or biologic therapy and any toxicity associated with these treatments has recovered to ≤ NCI-CTCAE Grade 1
10. At least 21 days must have elapsed prior to Day 1 Cycle 1 since radiotherapy (limited palliative radiation is allowed > 2 weeks), immunotherapy or following major surgery and any surgical incision should be completely healed

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Uncontrolled infection or systemic disease.
3. Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease, angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
4. Patients with QTc of > 470 msec on screening ECG. (If a patient has QTc interval >470 msec on screening ECG, the screening ECG may be repeated twice (at least 24 hours apart). The average QTc from the 3 screening ECGs must be <470 msec in order for the patient to be eligible for the study.
5. Any major surgery, radiotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed > 2 weeks).
6. Chemotherapy regimens with delayed toxicity within the last 4 weeks. Chemotherapy regimens given continuously or on a weekly basis with limited potential or delayed toxicity within the last 2 weeks.
7. No concurrent systemic chemotherapy or biologic therapy is allowed.
8. Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both).
9. History of solid organ transplantation.
10. Psychiatric disorder or social or geographic situation that would preclude study participation.
11. Known unsuitability for treatment with carboplatin including renal disease where there is impaired glomerular filtration rate (GFR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Kelly, Study Director — Noxopharm Limited
Locations (4):
- Georgia (4):
  - Academician Z.Tskhakaia West Georgia National Center of Interventional Medicine" LTD/ Oncology Unit- JSC "EVEX Medical Corporation" group member, Kutaisi
  - Tbilisi State Medical University's First University Clinic, Department Of Oncology, Tbilisi
  - LTD, Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
  - JSC, Neo Medi, Tbilisi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measure will be made available within 12 months after study completion
Supporting Information: Study Protocol, CSR
Time Frame: 12-18 months after study completion

RESULTS

PARTICIPANT FLOW:
Groups:
- NOX66 400 mg: NOX66 400 mg administered daily for 14 days in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
- NOX66 800 mg: NOX66 800 mg administered daily for 14 days in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
Period: Monotherapy
Arm/Group | NOX66 400 mg | NOX66 800 mg
Started | 8 (8 received NOX66 400 mg monotherapy and combination therapy with carboplatin.) | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Carboplatin Combination Therapy
Arm/Group | NOX66 400 mg | NOX66 800 mg
Started | 8 (All continued to combination therapy) | 10 (7 continued to combination therapy; 3 started combination therapy only)
Completed | 3 | 6
Not Completed | 5 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 2
Not completed — Disease progression | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled population = 19 Safety population includes those that received at least 1 NOX66 dose = 18 (n=8 in 400 mg arm; n=10 in 800 mg arm) Efficacy population = 14 (n=5 in 400 mg arm; n=9 in 800 mg arm)
Groups:
- Total: Total of all reporting groups
Arm/Group | NOX66 400 mg | NOX66 800 mg | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Georgia | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Dose Limiting Toxicity (DLT) During NOX66 Monotherapy and During NOX66 Combination With Carboplatin
Description: Dose limiting toxicity during monotherapy and combination therapy defined as any Grade 3 or more toxicity (by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE version 4.03]) (related to therapy) excluding Grade 3 or more neutropenia lasting greater than 5 days or thrombocytopenia associate with bleeding or Grade 4 thrombocytopenia.
Time Frame: Up to 1 month for NOX66 monotherapy from enrollment and up to 7 months from start of NOX66 combination therapy
Population: All participants that received at least one dose of NOX66; 3 participants in 800 mg group did not receive monotherapy
Measure: Count of Participants; unit: Participants
Groups:
- NOX66 400 mg Monotherapy: NOX66 400 mg administered daily for 14 days in a 21-day monotherapy (period 1)
- NOX66 400 mg Combination Therapy: NOX66 400 mg administered daily for 14 days in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
- NOX66 800 mg Monotherapy: NOX66 800 mg administered daily for 14 days in a 21-day monotherapy (period 1)
- NOX66 800 mg Combination Therapy: NOX66 800 mg administered daily for 14 days in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
Arm/Group | NOX66 400 mg Monotherapy | NOX66 400 mg Combination Therapy | NOX66 800 mg Monotherapy | NOX66 800 mg Combination Therapy
Number analyzed (Participants) | 8 | 8 | 7 | 10
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Treatment Emergent Adverse Events (SAEs) Related to NOX66.
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. Treatment-related are events which had causal relationship to study drug as assessed by the Investigator and were suspected to be reasonably related to the study drug.
Time Frame: From enrollment through 30 days after the last cycle of therapy (8 months)
Population: Safety analyses set included all enrolled participants who received at least 1 dose of NOX66 or 1 dose NOX66 and carboplatin.
Measure: Count of Participants; unit: Participants
Arm/Group | NOX66 400 mg Monotherapy | NOX66 400 mg Combination Therapy | NOX66 800 mg Monotherapy | NOX66 800 mg Combination Therapy
Number analyzed (Participants) | 8 | 8 | 7 | 10
Participants | 0 | 0 | 1 | 0

3. Secondary Outcome: Objective Response Rate (ORR) at Cycle 3 and at Cycle 6 of Combination Therapy
Description: Objective response rate defined as the percentage of participants achieving a complete response (CR) and or partial response (PR) after treatment with NOX66 and carboplatin therapy as assessed by Response Evaluation Criteria in solid tumors (RECIST) v1.1.
  CR defined as disappearance of all target and non-target lesions and reduction of any pathological lymph nodes (whether target or non-target) to <10 mm in short axis; PR was defined by a 30% or more decrease in sum of longest diameter (SLD) of target lesions in reference to baseline. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and no new lesions.
Time Frame: Radiological evaluation at baseline and at 3 months and at 6 months
Population: Participants with measurable disease by RECIST v1.1 criteria at baseline and at 3 and 6 month post start of combination therapy.
Measure: Count of Participants; unit: Participants
Groups:
- NOX66 400 mg + Carboplatin (AUC4) to Cycle 3: NOX66 400 mg administered daily for 14 day in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with low dose carboplatin AUC = 4 for treatment cycles 1-3
- NOX66 400 mg + Carboplatin (AUC6) to Cycle 6: NOX66 400 mg administered daily for 14 day in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
- NOX66 800 mg + Carboplatin (AUC4) to Cycle 3: NOX66 800 mg administered daily for 14 day in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with low dose carboplatin AUC = 4 for treatment cycles 1-3
- NOX66 800 mg + Carboplatin (AUC6) to Cycle 6: NOX66 800 mg administered daily for 14 day in a 21-day monotherapy (period 1) followed by 28-day combination therapy cycle (period 2) whereby NOX66 administered on days 1 to 7 and IV carboplatin on Day 2 in each cycle with 2 carboplatin doses low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
Arm/Group | NOX66 400 mg + Carboplatin (AUC4) to Cycle 3 | NOX66 400 mg + Carboplatin (AUC6) to Cycle 6 | NOX66 800 mg + Carboplatin (AUC4) to Cycle 3 | NOX66 800 mg + Carboplatin (AUC6) to Cycle 6
Number analyzed (Participants) | 5 | 2 | 9 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1

4. Secondary Outcome: Overall Clinical Response Rate at Cycle 3 and at Cycle 6 of Combination Therapy
Description: Overall Clinical response rate defined as the percentage of participants who achieved complete response (CR) or partial response (PR) or stable disease (SD) as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) criteria v1.1 after combination of NOX66 and carboplatin therapy.
  CR defined as disappearance of all target and non-target lesions and reduction of any pathological lymph nodes (whether target or non-target) to <10 mm in short axis; PR was defined by a 30% or more decrease in sum of longest diameter (SLD) of target lesions in reference to baseline. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD was defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Radiological evaluation at baseline and at 3 months and at 6 months
Population: Participants with evaluable (measurable ) disease by RECIST v1.1 criteria at baseline and at 3 month and 6 month post combination therapy
Measure: Count of Participants; unit: Participants
Arm/Group | NOX66 400 mg + Carboplatin (AUC4) to Cycle 3 | NOX66 400 mg + Carboplatin (AUC6) to Cycle 6 | NOX66 800 mg + Carboplatin (AUC4) to Cycle 3 | NOX66 800 mg + Carboplatin (AUC6) to Cycle 6
Number analyzed (Participants) | 5 | 2 | 9 | 6
Participants | 4 | 1 | 7 | 5

ADVERSE EVENTS:
Time Frame: 7 months
Groups:
- Monotherapy Phase, NOX66 400 mg: NOX66 400 mg administered daily for 14 day in a 21-day monotherapy phase (period 1)
- Monotherapy Phase, NOX66 800 mg: NOX66 800 mg administered daily for 14 day in a 21-day monotherapy phase (period 1)
- Combination Phase, NOX66 400 mg: Up to 6 cycles of a 28-day combination therapy cycle (period 2) with NOX66 400 mg administered daily on days 1 to 7 and IV carboplatin administered on Day 2 in each cycle with 2 carboplatin doses - low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
- Combination Phase, NOX66 800 mg: Up to 6 cycles of a 28-day combination therapy cycle (period 2) with NOX66 800 mg administered daily on days 1 to 7 and IV carboplatin administered on Day 2 in each cycle with 2 carboplatin doses - low dose carboplatin AUC = 4 for treatment cycles 1-3 followed by higher dose carboplatin AUC = 6 for treatment cycles 4-6.
Arm/Group | Monotherapy Phase, NOX66 400 mg | Monotherapy Phase, NOX66 800 mg | Combination Phase, NOX66 400 mg | Combination Phase, NOX66 800 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 1/8 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 1/8 | 3/10
Other Adverse Events (participants affected / at risk) | 1/8 | 1/7 | 6/8 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Monotherapy Phase, NOX66 400 mg (N=8) | Monotherapy Phase, NOX66 800 mg (N=7) | Combination Phase, NOX66 400 mg (N=8) | Combination Phase, NOX66 800 mg (N=10)
sudden death (General disorders) | 0 (0) | 0/3 (0) | 1 (1) | 0 (0) — sudden death
Infusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — related to carboplatin infusion
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — intestinal bleed
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy Phase, NOX66 400 mg (N=8) | Monotherapy Phase, NOX66 800 mg (N=7) | Combination Phase, NOX66 400 mg (N=8) | Combination Phase, NOX66 800 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (7)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy, peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism, arterial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to Phase 1 nature of the study, the subject sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT02941523/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02941523/SAP_001.pdf